CLINICAL TRIAL: NCT03800355
Title: An Observational, Retrospective Study on the Progress of Breast Cancer Cases in Males and the Assessment of Relapse Risk Through Gene Sequencing
Brief Title: Study on the Progress of Breast Cancer Cases in Males and the Assessment of Relapse Risk
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Fundación ADEY (Unknown)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2016-04
Record Dates: First submitted 2018-06-22; First posted 2019-01-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer, Male
Keywords: Breast Cancer in males; Observational; Gene Sequencing
MeSH Terms: conditions — Breast Neoplasms, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor tissue and blood samples will be collected and biological and genetic analyses will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male breast cancer: The study target population is all cases of male breast cancer (MBC), diagnosed with invasive breast cancer between the years 2000 and 2019, and treated in the Medical Oncology Departments of participating sites.

SUMMARY:
An observational, Other Designs (OD) post-marketing, multicenter study, which will obtain retrospective data from male patients diagnosed with invasive breast cancer between 2000 and 2019 in the medical oncology departments of hospitals that are associated with Spanish Breast Cancer Research Group (GEICAM) (using information obtained from patient medical histories).

DETAILED DESCRIPTION:
One of the objectives of this project is to ensure representativeness of the cases referred to. Accordingly, participating sites agree to enroll in the study male patients who were diagnosed with breast cancer in the period between 2000 and 2019.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with primary invasive breast carcinoma between the years 2000-2019, and who have been treated and/or followed up in the Medical Oncology Departments of participating sites.
* The enrollment of patients who died is allowed.

Exclusion Criteria:

* Male patients who do not wish to participate in the study for any reason.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study target population is all cases of male breast cancer (MBC), diagnosed with invasive breast cancer between the years 2000 and 2019, and treated in the Medical Oncology Departments of participating sites.
Sampling Method: Probability Sample
Enrollment: 777 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
General condition: Age | From date of patient breast cancer diagnosis until 2019.
  General condition age will be recorded.
General condition: performance status at diagnosis | From date of patient breast cancer diagnosis until 2019.
  Performance status by Eastern Cooperative Oncology Group (ECOG) Scale
General condition and history: substance abuse | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With Substance abuse of tobacco and alcohol will be recorded.
Diagnosis of other primary tumors | From date of patient breast cancer diagnosis until 2019.
  Diagnosis of other primary tumors synchronous or metachronous, will be recorded.
Body mass index (BMI) | From date of patient breast cancer diagnosis until 2019.
  BMI is a value derived from the mass (weight) and height. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Primary comorbidities | From date of patient breast cancer diagnosis until 2019.
  Primary comorbidities will be recorded.
Mutational status of BReast CAncer gene (BRCA) or other genes of genetic predisposition | From date of patient breast cancer diagnosis until 2019.
  Mutational status of BRCA or other genes of genetic predisposition will be recorded.
Family history of cancer | From date of patient breast cancer diagnosis until 2019.
  Family history of cancer will be recorded.
Anatomopathological characteristics of the tumor: date of diagnosis | From date of patient breast cancer diagnosis until 2019.
  Date of diagnosis will be collected.
Anatomopathological characteristics of the tumor: histology | From date of patient breast cancer diagnosis until 2019.
  The histology of the tumor will be collected
Anatomopathological characteristics of the tumor: clinical and/or pathological stage | From date of patient breast cancer diagnosis until 2019.
  Tumor clinical and/or pathological stage will be collected through the tumor-node-metastasis (TNM) staging system of the Union for International Cancer Control (UICC).
Anatomopathological characteristics of the tumor: hormone-receptor expression | From date of patient breast cancer diagnosis until 2019.
  Hormone-receptor expression will be collected
Anatomopathological characteristics of the tumor: Human Epidermal Growth Factor Receptor 2 (HER-2) expression | From date of patient breast cancer diagnosis until 2019.
  Human Epidermal Growth Factor Receptor 2 (HER-2) expression will be collected
Anatomopathological characteristics of the tumor: histologic grade | From date of patient breast cancer diagnosis until 2019.
  Tumor histologic grade will be collected
Anatomopathological characteristics of the tumor: Ki-67 | From date of patient breast cancer diagnosis until 2019.
  Tumor Ki-67 proliferation index will be collected
Anatomopathological characteristics of the tumor: lymphovascular invasion | From date of patient breast cancer diagnosis until 2017.
  Number of Participants With Presence of lymphovascular invasion will be collected
Treatment data: date of surgery | From date of patient breast cancer diagnosis until 2019.
  Will be collected date of surgery
Treatment data: type of surgery | From date of patient breast cancer diagnosis until 2019.
  Number of participants with each type of surgery: mastectomy or lumpectomy or quadrantectomy or lymphadenectomy or sentinel lymph node biopsy will be collected.
Treatment data: type of chemotherapy | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With neoadjuvant chemotherapy and adjuvant chemotherapy.
Treatment data: adjuvant radiotherapy | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With adjuvant radiotherapy
Treatment data: adjuvant hormonotherapy | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With hormonotherapy
Treatment data: other type of anti-cancer treatment | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With other type of anti-cancer treatment.
Follow-up data: relapse type | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With each relapse type: local, regional or distant
Follow-up data: site of metastatic disease | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With site of metastatic disease
Follow-up data: occurrence of other primary tumors | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With occurrence of other primary tumors whether or not of breast origin (in situ or invasive).
Follow-up data: current condition | From date of patient breast cancer diagnosis until 2019.
  The date of the last review and current clinical condition will be recorded.

SECONDARY OUTCOMES:
Biological and molecular characteristics analyzed in primary tumors: tumor subtypes | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With tumor subtypes, luminal profiles (e.g., luminal subtypes M1/M2, intrinsic subtypes)
Biological and molecular characteristics analyzed in primary tumors: risk groups | From date of patient breast cancer diagnosis until 2019.
  Number of Participants With risk groups on the reference of breast cancer in women, including morphological analyses and description of the clinical profile (e.g., morphological type, differentiation (histologic grade), Estrogen Receptor (ER), Progesterone Receptor (PgR), Human Epidermal growth factor Receptor 2 (HER2), Androgen Receptor (AR), Ki-67).
Date and cause of death | From date of patient breast cancer diagnosis until 2019.
  Date and cause of death, when applicable.
Disease-free survival (DFS). | From date of patient breast cancer diagnosis until 2019.
  DFS: it is defined as the time from date of initial breast cancer diagnosis to the date of the first documented relapse event (local, regional and/or distant) of the disease, second breast or non-breast primary tumor, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
Distant metastasis-free survival (DMFS). | From date of patient breast cancer diagnosis until 2019.
  DMFS: it is defined as the time from date of initial breast cancer diagnosis to the date of the first documented distant relapse, second invasive non-breast primary tumor, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
Progression-free survival (PFS). | From date of patient breast cancer diagnosis until 2019.
  PFS: it is defined as the time from the start date of a specific treatment to the documentation of disease progression on such treatment, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
Overall survival (OS). | From date of patient breast cancer diagnosis until 2019.
  OS: it is defined as the time from the date of initial breast cancer diagnosis to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Investigator, Study Director — Hospital Universitario Ramón y Cajal, Madrid, Spain; Chief Medical Investigator, Study Director — Fundación Onkologikoa, San Sebastián, Spain
Locations (54):
- Spain (54):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital General de Granollers, Granollers, Barcelona
  - Instituto Catalán de Oncología de L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Consorci Corporació Sànitari Parc Taulí, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Basurto, Bilbao, Bizcaia
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital General La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipúzcoa
  - Onkologikoa, Donostia / San Sebastian, Guipúzcoa
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario San Agustín, Avilés, Principality of Asturias
  - Hospital de Tortosa Verge de la Cinta, Tortosa, Tarragona
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus-Grupo Quirónsalud-Instituto Oncológico Dr. Rosell, Barcelona
  - Hospital Universitari Vall D´Hebrón, Barcelona
  - IDOC Centre Médic, Barcelona
  - Hospital Virgen de la Luz, Cuenca
  - Instituto Catalán de Oncología de Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - GenesisCare Madrid Hospital La Milagrosa, Madrid
  - Hospital Central de la Defensa Gómez Ulla, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Zarzuela, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Nuestra Señora De Candelaria, Santa Cruz de Tenerife
  - Hospital de Sant Pau i Santa Tecla, Tarragona
  - Hospital Universitario de Toledo, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Quirón Zaragoza, Zaragoza
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org